CLINICAL TRIAL: NCT07277985
Title: Comparison of the C-MAC D-Blade Videolaryngoscope and the Macintosh Laryngoscope for Postoperative Vocal Cord Assessment After Thyroidectomy
Brief Title: C-MAC D-Blade vs Macintosh for Postoperative Vocal Cord Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Sami Akbulut, Professor of Surgery, Inonu University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2022/115
Record Dates: First submitted 2025-12-01; First posted 2025-12-11 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Postoperative Vocal Cord Mobility; Recurrent Laryngeal Nerve Injury
Keywords: Thyroidectomy; Macintosh Laryngoscope; Videolaryngoscope; Airway Management; Vocal Cord Mobility; Recurrent Laryngeal Nerve
MeSH Terms: conditions — Recurrent Laryngeal Nerve Injuries

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned in a 1:1 ratio to either the C-MAC D-Blade videolaryngoscope group or the Macintosh laryngoscope group. Both groups were followed and evaluated in parallel throughout the study.
Who Masked: Participant, Care Provider
Masking Description: Randomization was performed by an anesthesiologist not involved in the study procedures, ensuring that the participant, care provider, and investigator remained masked to group assignment. The outcomes assessor was not masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- C-MAC D-Blade Videolaryngoscope (Experimental): Patients in this group were intubated using the C-MAC D-Blade videolaryngoscope to facilitate glottic visualization and to perform postoperative vocal cord mobility assessment.
  Interventions: Device: Videolaryngoscope (C-MAC D-Blade)
- Macintosh Laryngoscope (Active Comparator): Patients in this group were intubated with the traditional Macintosh direct laryngoscope, which was also used for postoperative assessment of vocal cord mobility.
  Interventions: Device: Direct Laryngoscope (Macintosh)

INTERVENTIONS:
Device: Videolaryngoscope (C-MAC D-Blade) — The C-MAC D-Blade videolaryngoscope was used to perform endotracheal intubation and to obtain a video-assisted view of the glottis. Its angulated blade design allows indirect visualization, providing improved glottic exposure during intubation and postoperative vocal cord mobility assessment
  Arms: C-MAC D-Blade Videolaryngoscope
Device: Direct Laryngoscope (Macintosh) — The Macintosh direct laryngoscope was used for endotracheal intubation with conventional direct visualization of the glottis. This standard laryngoscopic technique was also used for postoperative assessment of vocal cord mobility.
  Other Names: Direct Laryngoscope; Macintosh Blade
  Arms: Macintosh Laryngoscope

SUMMARY:
This study compares two different laryngoscopes-the C-MAC D-Blade videolaryngoscope and the Macintosh direct laryngoscope-for evaluating vocal cord mobility after thyroidectomy. Patients undergo standard anesthesia and intubation with one of the two devices. After surgery, vocal cord function is assessed to identify early postoperative vocal cord impairment. The study aims to determine whether videolaryngoscopy provides a more reliable and less traumatic method for postoperative vocal cord evaluation compared with the traditional Macintosh laryngoscope.

DETAILED DESCRIPTION:
This prospective randomized study evaluates two laryngoscopic techniques used during endotracheal intubation in patients undergoing thyroidectomy. The C-MAC D-Blade videolaryngoscope provides an angulated blade and video-assisted view of the glottis, while the Macintosh laryngoscope represents the traditional direct visualization method. Because postoperative vocal cord impairment is an important early indicator of potential recurrent laryngeal nerve injury after thyroidectomy, accurate assessment immediately after surgery is clinically valuable.

In this study, eligible patients were randomly assigned to intubation using either the C-MAC D-Blade videolaryngoscope or the Macintosh laryngoscope. All procedures were performed under standard anesthesia protocols by experienced anesthesiologists. After extubation and recovery, vocal cord mobility was evaluated using a standardized six-grade scoring system to assess postoperative vocal cord function.

The study compares intubation characteristics, glottic views, optimization maneuvers, hemodynamic responses, and postoperative vocal cord mobility between the two devices. The primary aim is to determine whether videolaryngoscopy offers a more reliable and less traumatic method for postoperative vocal cord evaluation. Secondary objectives include evaluating ease of intubation, maneuver requirements, and perioperative physiological responses. The findings may help guide device selection for airway management in thyroid surgery and improve early detection of recurrent laryngeal nerve dysfunction.

ELIGIBILITY:
Inclusion Criteria

* Age between 20 and 70 years.
* Height greater than 145 cm.
* Body mass index (BMI) between 20 and 35 kg/m².
* American Society of Anesthesiologists (ASA) physical status
* Scheduled for elective thyroid surgery under general anesthesia.

Exclusion Criteria

* Prior neck surgery or radiotherapy
* Large thyroid mass causing severe anatomical distortion.
* Mouth opening less than 4 cm.
* Short neck less than 6 cm in length.
* Limited head and neck mobility
* Unexpected difficult intubation.
* Known history of recurrent laryngeal nerve injury
* Presence of any neurological disorder.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2023-01-23 (Actual); Primary Completion 2023-05-26 (Actual); Study Completion 2023-05-26 (Actual)

PRIMARY OUTCOMES:
Postoperative Vocal Cord Mobility Score | Within 30 minutes after extubation
  Vocal cord mobility will be assessed using a standardized six-grade scoring system (I-VI) to detect postoperative vocal cord impairment after thyroidectomy.

SECONDARY OUTCOMES:
Glottic View (Cormack-Lehane Grade) | During intubation procedure
  The view of the glottis during intubation will be assessed using the Cormack-Lehane grading system.
Need for Optimization Maneuvers | During intubation procedure
  Whether external laryngeal maneuvers or additional attempts were required to facilitate intubation.

CONTACTS AND LOCATIONS:
Locations (1):
- Inonu University, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because the dataset contains identifiable clinical information and the study was not designed with external data distribution in mind

REFERENCES:
- [Result] Chilkoti GT, Gupta A, Bhandari P, Mohta M. Techniques of detecting recurrent laryngeal nerve palsy in patients undergoing thyroid surgery: Pearls and pitfalls. J Anaesthesiol Clin Pharmacol. 2024 Apr-Jun;40(2):199-205. doi: 10.4103/joacp.joacp_346_22. Epub 2024 Apr 8. PMID 38919442
- [Result] Sastre JA, Lopez T, Del Barrio ME. Airtraq(R) videolaryngoscope for assessing vocal cord mobility at the end of thyroidectomy. J Clin Anesth. 2017 May;38:3-4. doi: 10.1016/j.jclinane.2017.01.012. Epub 2017 Jan 12. No abstract available. PMID 28372672
- [Result] Priyanka AS, Nag K, Hemanth Kumar VR, Singh DR, Kumar S, Sivashanmugam T. Comparison of King Vision and Truview Laryngoscope for Postextubation Visualization of Vocal Cord Mobility in Patients Undergoing Thyroid and Major Neck Surgeries: A Randomized Clinical Trial. Anesth Essays Res. 2017 Jan-Mar;11(1):238-242. doi: 10.4103/0259-1162.200240. PMID 28298792
- [Result] Kundra P, Kumar V, Srinivasan K, Gopalakrishnan S, Krishnappa S. Laryngoscopic techniques to assess vocal cord mobility following thyroid surgery. ANZ J Surg. 2010 Nov;80(11):817-21. doi: 10.1111/j.1445-2197.2010.05441.x. Epub 2010 Aug 19. PMID 20969690
- [Result] Chilkoti GT, Bhandari P, Mohta M, Saxena AK, Kapoor R. Comparison of the Efficacy of Macintosh Laryngoscope Versus Airtraq Videolaryngoscope for Visualization of Laryngeal Structures at the End of Thyroidectomy: A Randomized Control Study. Indian J Otolaryngol Head Neck Surg. 2023 Dec;75(4):3191-3198. doi: 10.1007/s12070-023-03828-9. Epub 2023 Jun 15. PMID 37974697
- [Result] Gangappa RB, Kenchannavar MB, Chowdary PB, Patanki AM, Ishwar M. Total Thyroidectomy for Benign Thyroid Diseases: What is the Price to be Paid? J Clin Diagn Res. 2016 Jun;10(6):PC04-7. doi: 10.7860/JCDR/2016/18733.7991. Epub 2016 Jun 1. PMID 27504342
- [Result] AlOsaif ZA, Al Bisher HM, Elshnawie HA, Al-Hariri MT. The Impact of Thyroidectomy and Lobectomy on Patients' Health-Related Quality of Life, Eastern Region, Saudi Arabia. Clin Pract. 2024 Jun 29;14(4):1251-1263. doi: 10.3390/clinpract14040101. PMID 39051295